CLINICAL TRIAL: NCT00356447
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study Investigating the Efficacy and Tolerability of Angeliq® (Drospirenone 2mg and Estradiol 1mg) in Postmenopausal Chinese Women With Vasomotor Symptoms Over Four 28-day Treatment Cycles.
Brief Title: Safety/Efficacy Study of Drospirenone/Estradiol to Treat Postmenopausal Chinese Women With Vasomotor Symptoms.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91442; 309341 (Other: Company internal)
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Vasomotor Symptoms
MeSH Terms: interventions — estradiol-drospirenone combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: Estradiol/DRSP (Angeliq, BAY86-4891)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estradiol/DRSP (Angeliq, BAY86-4891) — Drospirenone (DRSP) 2mg and Estradiol 1mg. One cycle consists of 28 days. One tablet daily for 28 days given for a total of 4 cycles. Oral administration.
  Arms: Arm 1
Drug: Placebo — Same administration.
  Arms: Arm 2

SUMMARY:
The study evaluates in Chinese post-menopausal women the combination of drospirenone 2 mg and estradiol 1 mg for the treatment of climacteric symptoms, such as hot flushes (vasomotor symptoms) and uro-genital complaints.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer HealthCare AG, Germany. Bayer HealthCare AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Chinese postmenopausal women with moderate to severe vasomotor symptoms

Exclusion Criteria:

* History of steroid hormone dependent malignant disease
* Known or suspected malignant or premalignant disease
* Current or history of severe heart, liver, renal, psychiatric disease
* Hyperlipemia

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2006-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Frequency of hot flushes | From baseline to week 16
Change in intensity of hot flushes | From baseline to week 16

SECONDARY OUTCOMES:
Change in other climacteric symptoms | From baseline to week 16
Vaginal Bleeding pattern | From baseline to week 16
Global clinical impression | From baseline to week 16

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- China (6):
  - Wuhan, Hubei
  - Nanjing, Jiangsu
  - Jinan, Shandong
  - Beijing
  - Chongqing
  - Shanghai